CLINICAL TRIAL: NCT02400099
Title: Protein-rich Diet and Non-Alcoholic Fatty Liver Disease in Bariatric Surgery
Brief Title: Protein-rich Diet and NAFLD in Bariatric Surgery
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Catholic University of the Sacred Heart (Other)
Collaborators: Federico II University (Other)
Responsible Party: Principal Investigator, Geltrude Mingrone, Associate Professor, Catholic University of the Sacred Heart
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: UCSC-2015
Record Dates: First submitted 2015-03-23; First posted 2015-03-26 (Estimated); Last update posted 2015-03-26 (Estimated); Status verified 2015-03

CONDITIONS: Obesity; Non-alcoholic Fatty Liver Disease
MeSH Terms: conditions — Obesity; Non-alcoholic Fatty Liver Disease | interventions — Body Composition; Metabolome

STUDY DESIGN:
Who Masked: Outcomes Assessor

ARMS (2):
- High-protein low calorie diet (HPLC) (Active Comparator): 900 Kcal; Protein 90 g (39%); CHO 75 g (30%); Lipid 32 g (31%)
  Interventions: Dietary Supplement: High-protein low calorie diet; Other: Anthropometrical measurements; Other: Body composition; Other: 8-h metabolic profile; Other: Liver biopsy
- Control low calorie diet (CLC) (Placebo Comparator): 900 Kcal; Protein. 50 g (22%); CHO 119 g (48%); Lipid 31 g (30%)
  Interventions: Dietary Supplement: Control low calorie diet; Other: Anthropometrical measurements; Other: Body composition; Other: 8-h metabolic profile; Other: Liver biopsy

INTERVENTIONS:
Dietary Supplement: High-protein low calorie diet
  Arms: High-protein low calorie diet (HPLC)
Dietary Supplement: Control low calorie diet
  Arms: Control low calorie diet (CLC)
Other: Anthropometrical measurements
Other: Body composition
Other: 8-h metabolic profile
Other: Liver biopsy

SUMMARY:
Randomized, single-blind, trial to determine whether a high-protein, low calorie diet is more effective than a control low calorie diet in improving the metabolic and histologic abnormalities in patients with Non-alcoholic Fatty Liver Disease undergoing bariatric surgery.

ELIGIBILITY:
Inclusion Criteria:

* Morbidly obese subjects with a BMI >40 kg/m2 who are eligible for bariatric surgery and have accepted to undergo RYGB
* Weight stable for at least 6 months before the study (+/- 5 kg within the previous 6 months)
* Stable medication
* Provision of informed consent

Exclusion Criteria:

* Patients not eligible for laparoscopic RYGB
* Incapacity to give a valid informed consent or unwilling to give the consent
* Pregnancy or lactating
* Type 2-diabetes mellitus
* Significant illness within the two weeks preceding surgery, as judged by the physician.
* Obvious infection (bacteria, virus etc)
* Major cardiovascular disease
* Major gastrointestinal, respiratory, or any hormonal disorders
* History of drug addiction and/or alcohol use
* Suspected or confirmed poor compliance
* Alcohol consumption of > 20 g per day in the case of women and > 30 g per day in the case of men for at least 3 consecutive months during the previous 5 years
* Presence of hepatitis C or frank cirrhosis.

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2015-06; Primary Completion 2016-06 (Estimated)

PRIMARY OUTCOMES:
Liver fat content assessment | 1 year

SECONDARY OUTCOMES:
Insulin sensitivity assessment | 1 year
fat free mass assessment | 1 year

CONTACTS AND LOCATIONS:
Locations (1):
- Catholic University School of Medicine, Rome, Italy